CLINICAL TRIAL: NCT05240326
Title: Investigation of the Effect of Clinical Pilates Training on Functional Exercise Capacity and Respiratory Muscle Performance in Patients With Rheumatoid Arthritis
Brief Title: The Effects of Pilates Training on Exercise Capacity and Respiratory Muscle Performance in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Selin Bayram, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-730
Record Dates: First submitted 2022-02-05; First posted 2022-02-15 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; respiratory muscle strength; respiratory muscle endurance; exercise capacity
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise training group (Active Comparator): Clinical pilates exercises
  Interventions: Other: exercise training group
- control training group (Sham Comparator): Relaxation exercises
  Interventions: Other: control training group

INTERVENTIONS:
Other: exercise training group — All exercise program will be applied during supervised session by a physiotherapist. Clinical pilates exercises will be performed three days in a week. Treatment will continue an hour in per session for 8 weeks. The program consisted of 10 minutes warm-up exercises, clinical pilates-based exercises on mat for 40 minutes and 10 minutes relaxation and stretching exercises.
  Arms: exercise training group
Other: control training group — The control group will be followed up as a home program by giving the relaxation exercises. Patients will be asked to do the exercises regularly for 3 days/week, 1 sessions/day, for eight weeks. Patients in the control group will be followed up by phone once a week.
  Arms: control training group

SUMMARY:
Rheumatoid arthritis (RA) is a chronic inflammatory disease associated with significant functional impairment and increased risk for cardiovascular and pulmonary disease. Along with pharmacological therapy, exercise seems to be a very promising intervention to improve disease-related outcomes, including functional capacity and systemic manifestations. Despite the fact that aerobic and strengthening exercises have been shown to be useful in patients with RA, there have been limited research on the effects of pilates training. Therefore, we aimed to investigate the effect of clinical pilates training on exercise capacity, respiratory and peripheral muscle strength, respiratory muscle endurance, respiratory function, pain, balance, core stability, dyspnea, functional status, fatigue, quality of life, depression and anxiety in patients with RA.

DETAILED DESCRIPTION:
According to sample size calculation 30 patients with RA will be included. Patients will be evaluated before and after treatment. Patients will be randomized into exercise and control training groups. In the exercise training group the patients will be given pilates exercise; in the control training group, the patients will be given relaxation exercise. Pilates exercises will be applied by the physiotherapist 3 days a week for 8 weeks. The patients in the control training group will be given relaxation exercises as a home exercise program 3 days a week for 8 weeks. Exercise capacity, pulmonary functions, respiratory and peripheral muscle strength, respiratory muscle endurance, pain, balance, core stability, dyspnea, functional status, fatigue, quality of life, depression and anxiety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Being diagnosed according to the American College of Rheumatology (ACR)/EULAR 2010 rheumatoid arthritis diagnostic criteria
* under standard medications

Exclusion Criteria:

* orthopedic or neurological disease with a potential to affect functional capacity
* have problems that can prevent evaluation
* have a neurological problem that may cause hearing or vision impairment
* changes in medical treatment in the last 3 months
* have high disease activity score (DAS-28>3.2)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength | First day
  Maximal inspiratory and expiratory muscle strength will be evaluated using mouth pressure device.
Respiratory muscle endurance | First day
  It will be assessed using an incremental threshold loading test, in which patients began with a load of 30% of maximum inspiratory pressure and increased by 10% every 2 minutes.
Functional exercise capacity | First day
  It will be evaluated with 6-minute walking test according to the American Thoracic Society and European Respiratory Society criteria.
Pulmonary functions contains dynamic lung volumes | First day
  Spirometry will be used to perform pulmonary function testing in accordance with the American Thoracic Society and European Respiratory Society guidelines.

SECONDARY OUTCOMES:
Peripheral muscle strength | Second day
  Upper and lower extremity muscle strength using portable hand held dynamometer, hand grip strength using grip dynamometer will be evaluated.
Pain level | First day
  It will be assessed using with Visual Analog Scale (VAS). VAS is a scale which consists of a 100-millimetre scale ranging from 0 (no pain at all) to 100 (worst imaginable pain). A higher score indicates greater pain intensity.
Balance | Second day
  The "Biodex Balance System®" will be used to test static balance. As a consequence of the test, the system will provide the general stability index, anterior/posterior (AP) stability index, medial/lateral (ML) stability index, and their standard deviations.
Core stability | Second day
  "Core" endurance and "core" power are the specific components of "core" stability and will be evaluated separately. Core muscle endurance times will assessed by using trunk extension, trunk flexion, and side bridge tests. Core power will assessed by using sit-ups ve modified push-ups tests.
Dyspnea | First day
  The Modified Medical Research Council (MMRC) dyspnea scale will be used to determine the perception of dyspnea during activities of daily living.
  Dyspnea is graded as: zero (shortness of breath with strenuous exercise only); one (shortness of breath when rushing or walking up a slight uphill); two (because of shortness of breath they walk slower than people of the same age or have to stop to breathe while walking at their own pace); three (stops to breathe after walking 100 meters or after a few minutes); and four (too short of breath to leave the house or shortness of breath when getting dressed).
Functional status | First day
  Functional status will be assessed by Health Assessment Questionnaire (HAQ).
  HAQ consists of 20 questions, each question is scored between 0-3. A high score indicates poor functional status.
Fatigue | Second day
  Fatigue will be evaluated using Turkish version of Fatigue Severity Scale.
  This questionnaire includes 9 items and score range for each item from 1 to 7 point (7-point Likert scale). Fatigue Severity Scale score is calculates by deriving an arithmetic mean. Cut-scores of over 4 are indicative of significant fatigue (higher scores show more severe fatigue).
Disease Specific Quality of Life | Second day
  Quality of life will be evaluated using Turkish version of the Rheumatoid Arthritis Quality of Life (RAQoL) questionnaire.
  This questionnaire includes 30 items, each question is scored 0 (no) or 1 (yes). A high score indicates poor quality of life.
Anxiety and depression | Second day
  Anxiety and depression will be evaluated using Turkish version of Hospital Anxiety and Depression (HAD) scale.
  HAD scale uses to determine the risk group of patients in terms of anxiety ad depression and consists of 14 questions. Lowest score that patients can get from both subscales is 0, the highest score 21. The cut-off points for the Turkish version of the HAD scale were 10 for the anxiety subscale (HAD-A) and 7 for the depression subscale (HAD-D).

CONTACTS AND LOCATIONS:
Overall Officials: Deran Oskay, Prof, Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yentur SB, Atas N, Ozturk MA, Oskay D. Comparison of the effectiveness of pilates exercises, aerobic exercises, and pilates with aerobic exercises in patients with rheumatoid arthritis. Ir J Med Sci. 2021 Aug;190(3):1027-1034. doi: 10.1007/s11845-020-02412-2. Epub 2020 Oct 22. PMID 33094465
- [Background] Byrnes K, Wu PJ, Whillier S. Is Pilates an effective rehabilitation tool? A systematic review. J Bodyw Mov Ther. 2018 Jan;22(1):192-202. doi: 10.1016/j.jbmt.2017.04.008. Epub 2017 Apr 26. PMID 29332746
- [Background] Silva HJA, Lins CAA, Nobre TTX, de Sousa VPS, Caldas RTJ, de Souza MC. Mat Pilates and aquatic aerobic exercises for women with fibromyalgia: a protocol for a randomised controlled blind study. BMJ Open. 2019 Feb 19;9(2):e022306. doi: 10.1136/bmjopen-2018-022306. PMID 30782866
- [Background] Kucukdeveci AA. Nonpharmacological treatment in established rheumatoid arthritis. Best Pract Res Clin Rheumatol. 2019 Oct;33(5):101482. doi: 10.1016/j.berh.2019.101482. Epub 2020 Jan 25. PMID 31987686